CLINICAL TRIAL: NCT05881057
Title: Application of Surface-enhanced Raman Scatting (SERS) Technology Based Intraoperative Navigation System in Lung Cancer
Brief Title: Application of SERS Technology Based Intraoperative Navigation System in Lung Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Yayi He, Principal Investigator, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: 2022HY0519
Record Dates: First submitted 2023-05-19; First posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Lung Cancer
Keywords: surgical margin; PH; prognosis; mass-spectrometry; Surface-enhanced Raman Scatting (SERS)
MeSH Terms: conditions — Lung Neoplasms; Margins of Excision

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to explore the application of Surface-enhanced Raman Scatting (SERS) technology in lung cancer surgery and clarify its mechanism through multi-omics mass spectrometry platform, and then further prove the clinical transformation value of this technology.

DETAILED DESCRIPTION:
This study intends to apply the intraoperative navigation system based on Surface-enhanced Raman Scatting (SERS) technology to detect the PH of lung tissue, and to evaluate the benign and malignant resection margins of lung tissue based on this. In order to clarify the discrimination mechanism, a multi-omics mass spectrometry platform is planned to study the internal small molecules and pathway changes. In addition, the patients were followed up for five years to explore the correlation between the prognosis of patients and the PH of lung tissues and lymph nodes, which could prove the clinical transformation value of this technology.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in clinical research; Fully understand and informed the study and sign the informed consent form (ICF); Be willing to follow and be able to complete all trial procedures.
2. Male or female aged 18-75 years or more when signing ICF.
3. Extended tumor resection was performed to remove the lung tumor tissue, and the resection margin was ≥2cm from the tumor margin.
4. The effective measured diameter of all the lung tissues to be measured was greater than 0.5cm.
5. The patient had not received previous systemic therapy for cancer.

Exclusion Criteria:

1. Unresectable lung cancer patients.
2. Patients had received previous systemic therapy for lung cancer.
3. Patients with other active malignant tumors within the past year or at the same time.
4. The patient had a known history of psychotropic drug abuse or drug use; She had a history of alcohol abuse.
5. According to the investigator's judgment, the patient had other factors that may lead to the early termination of the study.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-small cell lung cancer surgery patients in Shanghai Pulmonary Hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Overall Survival(OS) | From date of randomization until the date of death from any cause, whichever came first, assessed up to 60 months
  Time from randomization to death (from any cause).
Recurrence free survival(RFS) | From date of randomization until the date of first documented progression from any cause, whichever came first, assessed up to 60 months
  The time from surgery to recurrence or the end of follow-up was defined.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] National Lung Screening Trial Research Team; Aberle DR, Adams AM, Berg CD, Black WC, Clapp JD, Fagerstrom RM, Gareen IF, Gatsonis C, Marcus PM, Sicks JD. Reduced lung-cancer mortality with low-dose computed tomographic screening. N Engl J Med. 2011 Aug 4;365(5):395-409. doi: 10.1056/NEJMoa1102873. Epub 2011 Jun 29. PMID 21714641
- [Result] Becker N, Motsch E, Trotter A, Heussel CP, Dienemann H, Schnabel PA, Kauczor HU, Maldonado SG, Miller AB, Kaaks R, Delorme S. Lung cancer mortality reduction by LDCT screening-Results from the randomized German LUSI trial. Int J Cancer. 2020 Mar 15;146(6):1503-1513. doi: 10.1002/ijc.32486. Epub 2019 Jun 20. PMID 31162856
- [Result] Pastorino U, Silva M, Sestini S, Sabia F, Boeri M, Cantarutti A, Sverzellati N, Sozzi G, Corrao G, Marchiano A. Prolonged lung cancer screening reduced 10-year mortality in the MILD trial: new confirmation of lung cancer screening efficacy. Ann Oncol. 2019 Oct 1;30(10):1672. doi: 10.1093/annonc/mdz169. No abstract available. PMID 31168572
- [Result] Edwards JG, Chansky K, Van Schil P, Nicholson AG, Boubia S, Brambilla E, Donington J, Galateau-Salle F, Hoffmann H, Infante M, Marino M, Marom EM, Nakajima J, Ostrowski M, Travis WD, Tsao MS, Yatabe Y, Giroux DJ, Shemanski L, Crowley J, Krasnik M, Asamura H, Rami-Porta R; International Association for the Study of Lung Cancer Staging and Prognostic Factors Committee, Advisory Board Members, and Participating Institutions. The IASLC Lung Cancer Staging Project: Analysis of Resection Margin Status and Proposals for Residual Tumor Descriptors for Non-Small Cell Lung Cancer. J Thorac Oncol. 2020 Mar;15(3):344-359. doi: 10.1016/j.jtho.2019.10.019. Epub 2019 Nov 13. PMID 31731014
- [Result] Saji H, Okada M, Tsuboi M, Nakajima R, Suzuki K, Aokage K, Aoki T, Okami J, Yoshino I, Ito H, Okumura N, Yamaguchi M, Ikeda N, Wakabayashi M, Nakamura K, Fukuda H, Nakamura S, Mitsudomi T, Watanabe SI, Asamura H; West Japan Oncology Group and Japan Clinical Oncology Group. Segmentectomy versus lobectomy in small-sized peripheral non-small-cell lung cancer (JCOG0802/WJOG4607L): a multicentre, open-label, phase 3, randomised, controlled, non-inferiority trial. Lancet. 2022 Apr 23;399(10335):1607-1617. doi: 10.1016/S0140-6736(21)02333-3. PMID 35461558
- [Result] Suzuki K, Watanabe SI, Wakabayashi M, Saji H, Aokage K, Moriya Y, Yoshino I, Tsuboi M, Nakamura S, Nakamura K, Mitsudomi T, Asamura H; West Japan Oncology Group and Japan Clinical Oncology Group. A single-arm study of sublobar resection for ground-glass opacity dominant peripheral lung cancer. J Thorac Cardiovasc Surg. 2022 Jan;163(1):289-301.e2. doi: 10.1016/j.jtcvs.2020.09.146. Epub 2020 Nov 12. PMID 33487427